CLINICAL TRIAL: NCT04571827
Title: The Influence of Expectations on Post-needling Soreness and Pain Processing After Dry Needling Treatment: an Experimental Study
Brief Title: The Influence of Expectations on Post-needling Soreness and Pain Processing After Dry Needling Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Eleuterio Atanasio Sánchez Romero, Professor Orofacial Pain AND Craniomandibular Disorders / Invasive Techniques in Physical Therapy / Orthopedic Manual Physical Therapist ( PT, MSc, PhD) International Doctorate, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Expectative Influence
Record Dates: First submitted 2020-08-30; First posted 2020-10-01 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Placebo Effect; Pain Intensity; Disability; Dry Needling
Keywords: placebo effect; Dry Needling; diffuse noxious inhibitory control; Myalgia
MeSH Terms: conditions — Pain; Myalgia | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Studio design:
  A randomized, longitudinal, experimental, prospective, parallel and double-blind clinical trial will be carried out in which both the study subject and the researcher who made the measurements do not know which treatment group they belong to.
  Participants The sample was composed of 42 healthy patients residing in the Community of Madrid, all of whom were personally recruited for the study. All of them will have 15 incisions with dry needles in the latent trigger point of the upper trapezium. All patients will read the information sheet that explains what the study will consist of, as well as the informed consent form, which they will voluntarily sign before the intervention.
  Each group will be given a different sentence: one group will attempt to influence with a positive expectation, another with a neutral expectation, and yet another will attempt to influence with a negative expectation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Before the treatment, it will be explained to the patient that the study seeks to observe if pain appears after the dry needling. During the explanation, the desired expectation will be introduced:
  * Group with positive expectation: "it is a very effective technique that achieves excellent results in the improvement of the cervical musculature"
  * Group with neutral expectations: "It's a physical therapy technique used to treat neck pain and we're investigating its effects"
  * Group with negative expectation: "this is a technique that will cause discomfort in the area of intervention of the cervical muscles after applying it ".
  Neither the subjects assigned to the groups nor the researchers who measured the variables knew which group they belonged to.
  Patients will be randomly assigned through GraphPad Software's QuickCals application (La Joya, CA, USA) to one of the 3 study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Effect (Experimental): Group with positive expectation: "it is a very effective technique that achieves excellent results in the improvement of the cervical musculature"
  Before the treatment, it will be explained to the patient that the study seeks to observe if pain appears after the dry needling. During the explanation, the desired expectation will be introduced.
  Interventions: Other: Dry Needling
- Nocebo Effect (Experimental): Group with negative expectation: "this is a technique that will cause discomfort in the area of intervention of the cervical muscles after applying it ".
  Before the treatment, it will be explained to the patient that the study seeks to observe if pain appears after the dry needling. During the explanation, the desired expectation will be introduced.
  Interventions: Other: Dry Needling
- Neutral Effect (Experimental): Group with neutral expectations: "It's a physical therapy technique used to treat neck pain and we're investigating its effects"
  Before the treatment, it will be explained to the patient that the study seeks to observe if pain appears after the dry needling. During the explanation, the desired expectation will be introduced.
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Dry Needling — Deep dry needling procedure
  All subjects received a deep dry neddling technique on a latent myofascial trigger point of the upper trapezius muscle by isolating it by a pincer grasp with the thumb and index finger. This myofascial trigger point was previously found following the diagnostic criteria described by Travell & Simons and Fernández-de-las-Peñas et al., and the deep dry needling intervention applied was based on the technique described by Hong.
  The patients were placed in a prone position. Prior to the technique, the area was disinfected with an antiseptic solution. Fifteen incisions were made with a 0.26x40mm monofilament needle. The number of local twitch response made were noted. After removing the needle, at the end a soft compression was made with a cotton to reduce the possible appearance of bleeding.

SUMMARY:
The general objective of the study is to determine the effectiveness on local mechanical hypoalgesia, pain intensity, disability and psychological variables of the deep dry needling technique on a latent trigger point of the upper trapezius muscle.

The specific objective of the study is to observe the interaction between patient expectations and hypoalgesic effects in patients who will receive the same technique but with different explanations about it before punction and which could influence on the modulation of post-punction pain.

DETAILED DESCRIPTION:
Study design:

A randomized, longitudinal, experimental, prospective, parallel and double-blind clinical trial was conducted, where both the study subject and the researcher performing the measurements do not know which treatment group they belong to.

Participants The sample was composed of 42 healthy patients residing in the Community of Madrid, all of whom were recruited personally for the study. All of them will have 15 incisions by dry needling in latent trigger point of the upper trapezium localized by palpation. All patients will read the information sheet explaining what the study will consist, as well as the informed consent form, which they will sign voluntarily beforehand. Patients were randomly assigned using GraphPad Software's QuickCals application (La Joya, CA, USA) to one of the 3 study groups.

Each group will be given a different sentence: one group will be attempted to influence with positive expectation, another with neutral expectation, and yet another will be attempted to influence with negative expectation.

Measurement instruments

Measurement of the range of movement by means of an inclinometer. To measure the range of movement the patient will be seated in a chair; feet supported on the floor, triple flexion of lower limbs of 90º (hip, knee and foot), back well supported and straight, head straight and look at the horizon. The inclinometer will be positioned to measure flexion, extension, right and left tilt and right and left rotation. The inclinometer for CROM (cervical range of motion) is approved and validated in different studies.

Measurement of pain threshold to pressure

A digital algometer was used to measure mechanical hyperalgesia. The model used was the X® brand, consisting of a 1 cm2 cylindrical rubber attached to a pressure gauge. It is calibrated in kilograms (kg) and pounds. The scale expressed in kg/cm2 was used. All patients were familiarized with this test through a trial session. They were instructed to say STOP when the pressure sensation changed to painful. Three perpendicular measurements were made on an active or latent myofascial trigger point situated in upper trapezium muscle, the mean was calculated and the data were recorded for analysis. A rest period of 30 seconds was established between the measurements. A dermographic pencil was used to mark these points prior to measurement. The intra-assay reliability is high in the upper trapezius muscle (ICC = 0.94-0.97). The minimum detectable change (CMD) for considering the results as clinically relevant in the upper trapezius fibres has been shown to be between 0.45 kgf and 1.13 kgf.

Procedural protocol

Prior to the technique, the patient will be explained that the study seeks to observe if pain appears after the dry needling procedure. During the explanation, the desired expectation will be introduced:

* Group with positive expectation: "it is a very effective technique that achieves excellent results in the improvement of the cervical musculature"
* Group with neutral expectations: "It's a physical therapy technique used to treat neck pain and we're investigating its effects"
* Group with negative expectation: "this is a technique that will cause discomfort in the area of intervention of the cervical muscles after applying it ".

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and X years of age.
* Presence of at least one latent myofascial trigger point in the upper trapezius muscle.
* Patients who speak and understand Spanish correctly.
* Subjects without previous experience in dry puncture treatment.

Exclusion Criteria:

* If patients had neurological signs and symptoms.
* Subjects with a history of trauma, fracture or previous spinal surgery.
* Subjects with a history of musculoskeletal and/or rheumatological diseases.
* Unsurpassed fear of needles
* Coagulation disorders
* Infiltration of corticosteroids or local anesthetics for one year prior to the study.
* Taking analgesic or anti-inflammatory medication the week before the study.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from base line, immediately after the intervention with dry needling; and 24 hours, 48 hours, 72 hours and 1 of week follow-up after the intervention with dry needling
  To evaluate the pain that the patient has, we use the VAS (Appendix 1). This is a 100 mm line that measures pain intensity. The left end of the line represents the absence of pain, while the right end represents the worst pain imaginable. The numerical pain intensity scale adds a numerical graduation where 1 is no pain and 10 is the worst pain imaginable. The confidence and reliability of this scale has been approved and validated in different studies. This scale will be used accompanying each CROM measurement as well as in pre-treatment measurements.

SECONDARY OUTCOMES:
Neck Disability Index | Change from base line, immediately after the intervention with dry needling; and 24 hours, 48 hours, 72 hours and 1 of week follow-up after the intervention with dry needling
  It will be used to measure the level of disability perceived by the patient as a result of their neck pain, after performing the technique and to check whether it appears during the control measurements. It is a questionnaire composed of 10 sections on different activities of daily living (ADLs); self-care, reading, lifting weights, driving, sleeping, recreational activities, work, concentration, pain intensity and headache. Each section scores from 0 to 5, with zero being no pain and five being the worst pain imaginable. (Maximum 50 points). Therefore, in order of appearance, of the 6 options, the first option of each item represents 0 and the last one 5. The higher the score obtained, the greater the patient's disability.
STAI (State-Trait Anxiety) | Change from base line, immediately after the intervention with dry needling; and 24 hours, 48 hours, 72 hours and 1 of week follow-up after the intervention with dry needling
  Questionnaire composed of 20 items with 4 points each that evaluate "state anxiety" (transitory emotional condition influenced by environmental factors that decrease or increase anxiety) and another 20 that evaluate "trait anxiety" (personality factor that predisposes to suffer or not suffer anxiety). The 2-part score ranks patients at a percentile to the general population. The higher the score, the greater the anxiety. It is one of the most widely used tools in research to measure levels of general anxiety.
Beck II (Depression) | Change from base line, immediately after the intervention with dry needling; and 24 hours, 48 hours, 72 hours and 1 of week follow-up after the intervention with dry needling
  A 21-item scale used to assess the severity of depression. The patient has to select for each item the response alternative that best reflects his/her state during the last week. The total score is obtained by adding up the values of the selected items, which range from 0 to 3. The commonly accepted cut-off points for grading intensity/severity are as follows: 0 to 9, no depression; 10 to 18, mild depression; 19 to 29, moderate depression, and ≥ 30 points, severe depression.
PCS (Pain Catastrophizing Scale) | Change from base line, immediately after the intervention with dry needling; and 24 hours, 48 hours, 72 hours and 1 of week follow-up after the intervention with dry needling
  It consists of 14 items valued on a 5-point scale. It evaluates the degree to which they have thoughts and feelings when they experience pain.
TSK (Tampa Scale for Kinesiophobia) | Change from base line, immediately after the intervention with dry needling; and 24 hours, 48 hours, 72 hours and 1 of week follow-up after the intervention with dry needling
  17 items, 4 points each where higher scores indicate higher levels of fear of movement.
PASS-20 (Pain Anxiety Symptoms Scale) | Change from base line, immediately after the intervention with dry needling; and 24 hours, 48 hours, 72 hours and 1 of week follow-up after the intervention with dry needling
  It has four 5-item subscales that measure avoidance, fearful thoughts, cognitive and physiological anxiety, and pain responses. Participants rate each item on a 6-point scale ranging from never (0) to always (5).
FPQ-III (Fear of Pain Questionnaire) | Change from base line, immediately after the intervention with dry needling; and 24 hours, 48 hours, 72 hours and 1 of week follow-up after the intervention with dry needling
  It consists of 30 items, each with 5 points that measure fear over specific situations that normally produce pain

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández Carnero, PhD, Study Director — Universidad Rey Juan Carlos; Eleuterio A Sánchez Romero, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Eleuterio A Sánchez, Madrid, Spain

REFERENCES:
- [Derived] Sanchez Romero EA, Lim T, Villafane JH, Boutin G, Riquelme Aguado V, Martin Pintado-Zugasti A, Alonso Perez JL, Fernandez Carnero J. The Influence of Verbal Suggestion on Post-Needling Soreness and Pain Processing after Dry Needling Treatment: An Experimental Study. Int J Environ Res Public Health. 2021 Apr 15;18(8):4206. doi: 10.3390/ijerph18084206. PMID 33921101